CLINICAL TRIAL: NCT01833546
Title: A Japanese Single Center, Open-label, Phase I Trial of TH-302 Given Intravenously to Subjects With Solid Tumors as Monotherapy or to Subjects With Advanced Pancreatic Cancer in Combination With Gemcitabine
Brief Title: A Japanese Phase 1 Trial of TH-302 in Subjects With Solid Tumors and Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200592-002
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumor; Pancreatic Cancer
Keywords: Solid tumor; Pancreatic cancer; TH-302; Gemcitabine; Evofosfamide
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — TH 302; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Evofosfamide 240 mg (Experimental)
  Interventions: Drug: Evofosfamide
- Evofosfamide 340 mg (Experimental)
  Interventions: Drug: Evofosfamide
- Evofosfamide 480 mg (Experimental)
  Interventions: Drug: Evofosfamide
- Evofosfamide 340 mg + Gemcitabine (Experimental)
  Interventions: Drug: Evofosfamide; Drug: Gemcitabine

INTERVENTIONS:
Drug: Evofosfamide — Evofosfamide infusion intravenously at an escalated dose of 240, 340 or 480 milligram per square meter (mg/m^2) on Day 1, 8 and 15 of each 28-day treatment cycle until progressive disease, unacceptable toxicity or withdrawal.
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 on Day 1, 8 and 15 of each 28-day treatment cycle until progressive disease, unacceptable toxicity or withdrawal.
  Arms: Evofosfamide 340 mg + Gemcitabine

SUMMARY:
This is a Japanese Phase 1, open-label, and dose-escalating trial of TH-302 as monotherapy in subjects with solid tumors and in combination with gemcitabine in subjects with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years of age
* Signed written informed consent form
* Histologically or cytologically confirmed advanced or metastatic solid tumor previously treated with one or more standard treatment regimen(s) or for which no effective therapy is available
* Histologically or cytologically confirmed locally advanced unresectable or metastatic pancreatic adenocarcinoma previously untreated with chemotherapy or systemic therapy
* Recovered from toxicities of prior anti-cancer treatment to Grade 1 or less
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* Acceptable liver function, renal function, hematologic status and coagulation status as defined in the protocol
* No clinically significant abnormalities in urinalysis
* Effective contraception for both male and female subjects if the risk of conception exists
* Other inclusion criteria apply

Exclusion Criteria:

* Prior anti-cancer treatment with more than 3 myelosuppressive cytotoxic chemotherapy regimens
* Prior treatment with gemcitabine for their advanced or metastatic pancreatic cancer, except for radiosensitizing doses of gemcitabine
* Prior radiotherapy to more than 30 percent of the bone marrow within 6 months prior to the trial entry
* Cardiac disease with New York Heart Association (NYHA) Class 3 or 4, within 6 months prior to the trial entry
* Clinically significant (that is, active) cardiovascular disease
* Seizure disorders requiring anticonvulsant therapy
* Known brain, leptomeningeal or epidural metastases (unless previously treated and well controlled for at least 3 months at the trial entry)
* Previously treated malignancies other than the current disease for at least 5 years at the trial entry
* Severe chronic obstructive or other pulmonary disease major surgery, within 4 weeks prior to the trial entry, without complete recovery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Anti-cancer treatment prior to trial entry
* Participation in an investigational drug or device trial within 4 weeks prior to the trial entry
* Known infection with human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C
* A history of allergic reactions
* Taking a medication that is either moderate or strong inhibitor or inducer of cytochrome P450 (CYP)3A4 or is a sensitive substrate of other cytochrome P450
* Pregnancy or lactation period
* Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial
* Unwillingness or inability to comply with the trial protocol for any reason
* Legal incapacity or limited legal capacity
* Other exclusion criteria apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2016-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Japan
Locations (2):
- Japan (2):
  - Research Site, Kashiwa
  - Research Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant (informed consent): 18 April 2013. Study completion date: 25 January 2016.
Groups:
- Evofosfamide 240 mg: Participants received evofosfamide infusion intravenously at a dose of 240 milligram per square meter (mg/m^2) on Day 1, 8 and 15 of each 28-day treatment cycle until progressive disease, unacceptable toxicity or participant withdrawal.
- Evofosfamide 340 mg: Participants received evofosfamide infusion intravenously at a dose of 340 mg/m^2 on Day 1, 8 and 15 of each 28-day treatment cycle until progressive disease, unacceptable toxicity or participant withdrawal.
- Evofosfamide 480 mg: Participants received evofosfamide infusion intravenously at a dose of 480 mg/m^2 on Day 1, 8 and 15 of each 28-day treatment cycle until progressive disease, unacceptable toxicity or participant withdrawal.
- Evofosfamide 340 mg + Gemcitabine: Participants received 340 mg/m^2 evofosfamide in combination with 1,000 mg/m^2 gemcitabine intravenously on Day 1, 8 and 15 of each 28-day treatment cycle until progressive disease, unacceptable toxicity or participant withdrawal.
Period: Overall Study
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Started | 3 | 3 | 8 | 6
Completed | 3 | 3 | 8 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all subjects who received at least 1 dose of the study drug (evofosfamide or gemcitabine).
Units Other Than Participants: Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine | Total
Number analyzed (Participants) | 3 | 3 | 8 | 6 | 20
Number analyzed (Subjects) | 3 | 3 | 8 | 6 | 20
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 65 years | 2 | 1 | 4 | 3 | 10
  Greater than or equal to (>=) 65 years | 1 | 2 | 4 | 3 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 5 | 1 | 8
  Male | 1 | 3 | 3 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Any Dose-Limiting Toxicity (DLT) During First Cycle - Day 1 to 28
Description: A DLT was defined as any of the following toxicities at any dose level that occurred during the first cycle, and were considered to be related to the study drug by the Investigator or the Sponsor: - Grade 3 or Grade 4 non-hematological toxicity, except for Grade 3 or Grade 4 nausea, vomiting and diarrhea, - Grade 3 or higher skin reactions or mucosal toxicities, - Febrile neutropenia, - Grade 3 alanine aminotransferase (ALT)/aspartate aminotransferase (AST) elevation lasting more than 7 days, - Grade 4 neutropenia lasting more than 5 days, - Grade 4 thrombocytopenia, - Grade 4 anemia, - Any non-preexisting Grade 2 or higher non-hematologic toxicity which, in the judgment of the Investigator and the Sponsor, was considered a DLT, - Any Grade 2 or higher non-hematologic toxicity that did not resolve to Grade 0 or Grade 1 toxicity by the start of the next cycle which, in the judgment of the Investigator and the Sponsor, was considered a DLT.
Time Frame: Day 1 up to Day 28 of Cycle 1
Population: The DLT Analysis Set included all participants who experienced a DLT during Cycle 1 or who did not experience a DLT, completed Cycle 1 and received 90% or more of all planned total dose of evofosfamide, and gemcitabine for the combination, during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 6 | 6
Participants | 0 | 0 | 1 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE), Serious TEAEs, TEAEs Leading to Death
Description: AE was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are events with start date on or after the date of first dose of study treatment and up to and including 30 days after the last dose of study treatment, or events with start date prior to the date of first dose of study treatment, and worsened in severity or become serious during treatment. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 33 months
Population: Safety population included all participants who received at least 1 dose of the study drug (evofosfamide or gemcitabine).
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Participants
  TEAEs | 3 | 3 | 8 | 6
  Serious TEAEs | 0 | 0 | 1 | 1
  TEAEs leading to death | 0 | 0 | 0 | 0

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Evofosfamide and Its Metabolite (Bromo-isophosphoramide Mustard [Br-IPM])
Time Frame: Monotherapy: pre-dose, 0.25, 0.5, 0.58, 0.75, 1, 1.08, 1.25, 1.5, 2, 2.5, 3.5, 4.5, 6.5, 8.5, 12.5 hours post-dose on Day 1 and 15; Combination therapy: pre-dose, 0.5, 0.66, 1, 2, 2.5, 3, 3.5, 4, 4.5, 6.5, 8, 10.5, 26.5 hours post-dose on Day 1 and 15
Population: The Pharmacokinetics (PK) Analysis Set included all participants who received at least 1 dose of evofosfamide (that is, actual total dose of evofosfamide > 0) and who provided sufficient data for a concentration-time profile for evofosfamide. Here "Number Analyzed" signifies those participants who were evaluated at the specified time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
hours
  Evofosfamide: Day 1 | 0.550 [0.25 to 0.70] | 0.250 [0.23 to 0.25] | 0.392 [0.25 to 0.57] | 0.550 [0.53 to 0.58]
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 0.22 [0.22 to 0.58] | 0.533 [0.25 to 0.55] | 0.267 [0.22 to 0.53] | 0.533 [0.52 to 0.55]
  Br-IPM: Day 1 | 0.550 [0.53 to 0.92] | 0.633 [0.58 to 1.02] | 0.575 [0.53 to 0.62] | 0.567 [0.53 to 0.98]
  Br-IPM: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Br-IPM: Day 15 | 0.600 [0.58 to 0.67] | 0.550 [0.53 to 0.68] | 0.567 [0.53 to 0.60] | 0.533 [0.52 to 0.55]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Gemcitabine and Its Metabolite (2',2'-Difluorodeoxyuridine [dFdU])
Description: Tmax was the time to peak concentration in plasma, obtained directly from the concentration versus time curve. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: The PK Analysis Set included all participants who received at least 1 dose of gemcitabine (that is, actual total dose of gemcitabine > 0) and who provided sufficient data for a concentration-time profile for gemcitabine. Here "Number Analyzed" signifies those participants who were evaluated at the specified time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
hours
  Gemcitabine: Day 1 | 0.500 [0.48 to 0.52]
  Gemcitabine: Day 15: number analyzed (Participants) | 3
  Gemcitabine: Day 15 | 0.500 [0.50 to 0.53]
  dFdU: Day 1 | 0.500 [0.48 to 0.52]
  dFdU: Day 15: number analyzed (Participants) | 3
  dFdU: Day 15 | 0.500 [0.50 to 0.53]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Evofosfamide and Its Metabolite (Bromo-isophosphoramide Mustard [Br-IPM])
Description: Maximum observed plasma concentration was assessed.
Time Frame: as for outcome 3
Population: The PK Analysis Set included all participants who received at least 1 dose of evofosfamide (that is, actual total dose of evofosfamide > 0) and who provided sufficient data for a concentration-time profile for evofosfamide. Here "Number Analyzed" signifies those participants who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Nanogram per milliliter (ng/mL)
  Evofosfamide: Day 1 | 6502.3 (29.8) | 10009.8 (8.4) | 14016.7 (14.5) | 9303.4 (7.2)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 7159.9 (5.3) | 10248.2 (5.9) | 14661.2 (9.9) | 8720.8 (12.8)
  Br-IPM: Day 1 | 63.37 (32.7) | 103.74 (64.8) | 224.95 (25.4) | 86.55 (58.3)
  Br-IPM: Day 15: number analyzed (Participants) | 3 | 3 | 6 | 3
  Br-IPM: Day 15 | 62.01 (30.7) | 149.36 (11.2) | 207.88 (22.0) | 124.92 (33.5)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Gemcitabine and Its Metabolite (2',2'-Difluorodeoxyuridine [dFdU])
Description: Maximum observed Plasma concentration was assessed. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
ng/mL
  Gemcitabine: Day 1 | 22596.2 (22.3)
  Gemcitabine: Day 15: number analyzed (Participants) | 3
  Gemcitabine: Day 15 | 21355.5 (4.0)
  dFdU: Day 1 | 33923.9 (23.1)
  dFdU: Day 15: number analyzed (Participants) | 3
  dFdU: Day 15 | 33631.4 (22.6)

7. Secondary Outcome: Terminal Rate Constant Associated With the Terminal Elimination Phase (λz) of Evofosfamide and Its Metabolite (Bromo-isophosphoramide Mustard [Br-IPM])
Description: Terminal rate constant was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 3
Population: The PK Analysis Set. Here "Number Analyzed" signifies those Participants who were evaluated at the specified time point. There were no Participants analyzed at certain time points (that is, Number Analyzed = 0) because there was no data collected for respective arms at those time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Per hour
  Evofosfamide: Day 1 | 1.012 (6.0) | 1.100 (12.3) | 1.094 (6.0) | 1.146 (10.3)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 1.007 (6.2) | 1.032 (2.5) | 0.951 (27.0) | 1.177 (6.0)
  Br-IPM: Day 1: number analyzed (Participants) | 1 | 1 | 8 | 0
  Br-IPM: Day 1 | 1.478 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 2.436 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 1.758 (18.8) |
  Br-IPM: Day 15: number analyzed (Participants) | 1 | 3 | 5 | 0
  Br-IPM: Day 15 | 1.669 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 2.701 (35.7) | 1.581 (19.5) |

8. Secondary Outcome: Terminal Rate Constant Associated With the Terminal Elimination Phase (λz) of Gemcitabine and Its Metabolite (2',2'-Difluorodeoxyuridine [dFdU])
Description: Terminal rate constant was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
Per hour
  Gemcitabine: Day 1: number analyzed (Participants) | 4
  Gemcitabine: Day 1 | 3.241 (9.6)
  Gemcitabine: Day 15: number analyzed (Participants) | 3
  Gemcitabine: Day 15 | 3.171 (9.9)
  dFdU: Day 1 | 0.0895 (45.4)
  dFdU: Day 15 | 0.0870 (54.0)

9. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Evofosfamide and Its Metabolite (Bromo-isophosphoramide Mustard [Br-IPM])
Description: Terminal half-life was calculated as ln(2)/λz. Where λz is a Terminal rate constant, which was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
hours
  Evofosfamide: Day 1 | 0.6850 (6.0) | 0.6304 (12.3) | 0.6334 (6.0) | 0.6049 (10.3)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 0.6881 (6.2) | 0.6716 (2.5) | 0.7285 (27.0) | 0.5889 (6.0)
  Br-IPM: Day 1: number analyzed (Participants) | 1 | 1 | 8 | 0
  Br-IPM: Day 1 | 0.4691 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 0.2846 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 0.3942 (18.8) |
  Br-IPM: Day 15: number analyzed (Participants) | 1 | 3 | 5 | 0
  Br-IPM: Day 15 | 0.4153 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 0.2566 (35.7) | 0.4384 (19.5) |

10. Secondary Outcome: Apparent Terminal Half-life (t1/2) of of Gemcitabine and Its Metabolite (2',2'-Difluorodeoxyuridine [dFdU])
Description: Terminal half-life was calculated as ln(2)/λz. Where λz is a Terminal rate constant, which was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
hours
  Gemcitabine: Day 1: number analyzed (Participants) | 4
  Gemcitabine: Day 1 | 0.2139 (9.6)
  Gemcitabine: Day 15: number analyzed (Participants) | 3
  Gemcitabine: Day 15 | 0.2186 (9.9)
  dFdU: Day 1 | 7.741 (45.4)
  dFdU: Day 15 | 7.964 (54.0)

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Sampling Time With Concentration at or Above the Lower Limit of Quantitation (AUC[0-t]) of Evofosfamide and Its Metabolite (Bromo-isophosphoramide Mustard [Br-IPM])
Description: Area under the concentration-time curve from time 0 to the last quantifiable concentration was assessed.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour per mL (ng*hour/mL)
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
ng*hour per mL (ng*hour/mL)
  Evofosfamide: Day 1 | 5266.9 (8.3) | 7864.2 (13.0) | 10416.1 (14.4) | 5989.5 (11.5)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 5232.4 (2.4) | 8191.1 (17.8) | 10742.8 (16.7) | 5616.4 (21.0)
  Br-IPM: Day 1 | 38.1 (41.1) | 61.7 (84.4) | 153.8 (25.0) | 47.7 (66.5)
  Br-IPM: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Br-IPM: Day 15 | 41.4 (24.3) | 101.2 (18.6) | 149.4 (23.6) | 77.0 (23.6)

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Sampling Time With Concentration at or Above the Lower Limit of Quantitation (AUC[0-t]) of Gemcitabine and Its Metabolite (2',2'-Difluorodeoxyuridine [dFdU])
Description: Area under the concentration-time curve from time 0 to the last quantifiable concentration was assessed. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
ng*hour/mL
  Gemcitabine: Day 1 | 10001.2 (21.8)
  Gemcitabine: Day 15: number analyzed (Participants) | 3
  Gemcitabine: Day 15 | 9576.0 (7.2)
  dFdU: Day 1 | 139397.1 (25.1)
  dFdU: Day 15: number analyzed (Participants) | 3
  dFdU: Day 15 | 116487.7 (28.6)

13. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC [0-infinity]) of Evofosfamide and Its Metabolite (Bromo-isophosphoramide Mustard [Br-IPM])
Description: Area under the concentration-time curve from time zero extrapolated to infinity, calculated as AUC(0-last) + last observed concentration (Clast)/terminal rate constant (λz), using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations. Where AUC(0-last) is area under the concentration-time curve from time 0 to the last quantifiable concentration was assessed. λz was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
ng*hour/mL
  Evofosfamide: Day 1 | 5296.2 (8.2) | 7904.7 (13.2) | 10459.6 (14.5) | 6049.5 (11.9)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 5261.3 (2.4) | 8233.3 (18.0) | 10786.6 (16.8) | 5664.9 (21.3)
  Br-IPM: Day 1: number analyzed (Participants) | 1 | 1 | 8 | 0
  Br-IPM: Day 1 | 90 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 105 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 174.6 (21.9) |
  Br-IPM: Day 15: number analyzed (Participants) | 1 | 3 | 5 | 0
  Br-IPM: Day 15 | 51 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 participant analyzed in this reporting group. | 115.1 (17.2) | 171.8 (16.8) |

14. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC [0-infinity]) of Gemcitabine and Its Metabolite (2',2'-Difluorodeoxyuridine [dFdU])
Description: Area under the concentration-time curve from time zero extrapolated to infinity, calculated as AUC(0-last) + last observed concentration (Clast)/terminal rate constant (λz), using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations. Where AUC(0-last) is area under the concentration-time curve from time 0 to the last quantifiable concentration was assessed. λz was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
ng*hour/mL
  Gemcitabine: Day 1: number analyzed (Participants) | 4
  Gemcitabine: Day 1 | 10719.5 (24.5)
  Gemcitabine: Day 15: number analyzed (Participants) | 2
  Gemcitabine: Day 15 | 9996.0 (1.3)
  dFdU: Day 1 | 159014.1 (35.3)
  dFdU: Day 15: number analyzed (Participants) | 3
  dFdU: Day 15 | 133203.0 (46.3)

15. Secondary Outcome: Apparent Total Body Clearance of (CL) of Evofosfamide
Description: Apparent total clearance (CL/F) was calculated as dose divided by area under the plasma concentration-time profile from time zero extrapolated to infinity (AUC[inf]).
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour per square meter
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Liter per hour per square meter
  Evofosfamide: Day 1 | 45.83 (8.0) | 43.05 (13.1) | 46.07 (14.6) | 56.23 (11.8)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 45.74 (1.5) | 41.74 (18.0) | 44.59 (17.7) | 60.43 (21.0)

16. Secondary Outcome: Apparent Total Body Clearance of (CL) of Gemcitabine
Description: Apparent total clearance (CL/F) was calculated as dose divided by area under the plasma concentration-time profile from time zero extrapolated to infinity (AUC[inf]). This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour per square meter
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
Liter per hour per square meter
  Gemcitabine: Day 1: number analyzed (Participants) | 4
  Gemcitabine: Day 1 | 93.29 (24.5)
  Gemcitabine: Day 15: number analyzed (Participants) | 2
  Gemcitabine: Day 15 | 101.04 (1.9)

17. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of Evofosfamide
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) was the apparent volume of distribution at steady-state.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per square meter
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Liter per square meter
  Evofosfamide: Day 1 | 21.71 (15.0) | 21.54 (2.4) | 21.79 (15.2) | 39.03 (7.1)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 20.26 (16.4) | 18.83 (9.6) | 21.35 (5.2) | 41.55 (9.0)

18. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of Gemcitabine
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) was the apparent volume of distribution at steady-state. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per square meter
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
Liter per square meter
  Gemcitabine: Day 1: number analyzed (Participants) | 4
  Gemcitabine: Day 1 | 34.41 (21.9)
  Gemcitabine: Day 15: number analyzed (Participants) | 2
  Gemcitabine: Day 15 | 43.71 (18.3)

19. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) of Evofosfamide
Description: Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by elimination rate constant [λz]) following single dose. Area under the plasma concentration-time curve from time zero to infinity, calculated (AUC0-inf) as AUC0-t + AUCextra. AUCextra represents an extrapolated value obtained by Clast / λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured plasma concentration is at or above lower limit of quantification (LLQ) and λz is the elimination rate constant. And the elimination rate constant obtained from linear regression of the terminal phase of the log transformed concentration-time data.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per square meter
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Liter per square meter
  Evofosfamide: Day 1 | 44.85 (10.3) | 39.16 (1.2) | 42.10 (15.3) | 49.07 (11.4)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 45.41 (5.3) | 40.44 (17.5) | 46.86 (19.5) | 51.34 (17.3)

20. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) of Gemcitabine
Description: Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by elimination rate constant [λz]) following single dose. Area under the plasma concentration-time curve from time zero to infinity, calculated (AUC0-inf) as AUC0-t + AUCextra. AUCextra represents an extrapolated value obtained by Clast / λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured plasma concentration is at or above lower limit of quantification (LLQ) and λz is the elimination rate constant. And the elimination rate constant obtained from linear regression of the terminal phase of the log transformed concentration-time data. This outcome was applicable for only combination arm in which evofosfamide was administered along with gemcitabine.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per square meter
Arm/Group | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 6
Liter per square meter
  Gemcitabine: Day 1: number analyzed (Participants) | 4
  Gemcitabine: Day 1 | 28.78 (29.8)
  Gemcitabine: Day 15: number analyzed (Participants) | 2
  Gemcitabine: Day 15 | 30.14 (1.2)

21. Secondary Outcome: Cumulative Amount of Evofosfamide Excreted From Time Zero to Time After Dosing (Ae0-t)
Description: Cumulative amount excreted in urine from time zero to the end of the last measurable concentration was reported.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram per square meter
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
milligram per square meter
  Evofosfamide: Day 1 | 22.913 (43.6) | 17.135 (66.6) | 38.771 (33.3) | 22.691 (82.0)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 11.674 (139.2) | 22.605 (53.7) | 40.049 (66.0) | 30.025 (31.6)

22. Secondary Outcome: Renal Clearance (CL) for Evofosfamide
Description: Renal clearance is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour per square meter
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Liter per hour per square meter
  Evofosfamide: Day 1 | 4.35 (41.4) | 2.18 (59.9) | 3.72 (34.4) | 3.79 (81.4)
  Evofosfamide: Day 15: number analyzed (Participants) | 3 | 3 | 5 | 3
  Evofosfamide: Day 15 | 2.23 (137.0) | 2.76 (76.4) | 3.73 (83.1) | 5.35 (15.4)

23. Secondary Outcome: Best Overall Response (BOR)
Description: BOR was determined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). BOR was defined as the best response of any of the confirmed complete response (CR), confirmed partial response (PR), stable disease (SD) and progressive disease (PD). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)=Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD was defined as at least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Number of participants with CR, PR, SD and PD were reported.
Time Frame: Time from first treatment to final assessment at 33 months
Population: Efficacy Analysis Set included all participants who received at least 1 planned dose of evofosfamide and who had a baseline tumor assessment and at least 1 tumor assessment according to RECIST version 1.1 after the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 0 | 0 | 2 | 2
  Progressive Disease | 2 | 3 | 4 | 3

24. Secondary Outcome: Number of Participants With Objective Response
Description: OR was determined according to RECIST v1.1. Objective response is defined as a best overall response of confirmed complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Number of participants with OR were reported.
Time Frame: Time from first treatment to final assessment at 33 months
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Participants | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Disease Control
Description: Disease Control was defined as having achieved at least disease stabilization; that is participants with confirmed CR, PR, or SD lasting for at least 16 weeks. CR: Disappearance of all target lesions. PR: A decrease of at least 30% in the sum of the longest diameter of target lesions. PD: PD is defined as at least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. SD: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: Time from first treatment to final assessment at 33 months
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Participants | 0 | 0 | 2 | 2

26. Secondary Outcome: Number of Participants With Clinical Significant Laboratory Abnormalities and Vital Signs Abnormalities Reported as Treatment Emergent Adverse Events
Description: Clinical laboratory parameters that were assessed included: hematological parameters, blood chemistry parameters, coagulation and urinalysis and the vital signs that were assessed included: blood pressure, heart rate, respiratory rate, and body temperature.
Time Frame: Baseline up to 33 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Participants
  Subjects with Lab Abnormalities | 3 | 3 | 8 | 6
  Subjects with Vital signs Abnormalities | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Twelve-lead ECGs were performed and assessed after at least 5 minutes rest in supine position locally.
Time Frame: Baseline up to 33 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Participants | 0 | 0 | 3 | 1

28. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 2 or Higher Than 2
Description: ECOG performance status measured to assess subject's performance status on a scale of 0 to 5, where 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (more than 50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=Death. Number of participants with ECOG performance status score of 2 or higher than 2 were reported.
Time Frame: Baseline up to 33 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
Number analyzed (Participants) | 3 | 3 | 8 | 6
Participants | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 33 months
Arm/Group | Evofosfamide 240 mg | Evofosfamide 340 mg | Evofosfamide 480 mg | Evofosfamide 340 mg + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/8 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evofosfamide 240 mg (N=3) | Evofosfamide 340 mg (N=3) | Evofosfamide 480 mg (N=8) | Evofosfamide 340 mg + Gemcitabine (N=6)
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Evofosfamide 240 mg (N=3) | Evofosfamide 340 mg (N=3) | Evofosfamide 480 mg (N=8) | Evofosfamide 340 mg + Gemcitabine (N=6)
Constipation (Gastrointestinal disorders) | 0 | 2 | 6 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Electrocardiogram QT Prolonged (Investigations) | 0 | 1 | 2 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 1 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 2 | 1
Neutrophil Count Decreased (Investigations) | 0 | 0 | 3 | 5
Blood Cholesterol Increased (Investigations) | 0 | 0 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 2 | 5
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 4
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 2
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 2 | 3
Pyrexia (General disorders) | 0 | 1 | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 3 | 1 | 3
Flushing (Vascular disorders) | 0 | 2 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0/6 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Tension Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 5
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other